CLINICAL TRIAL: NCT05518734
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple-dose Escalation Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of VX-708 in Healthy Subjects
Brief Title: A Phase 1 Dose Escalation Study of VX-708 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX22-708-003
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Itraconazole; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: VX-708 (Cohort A1-A3) (Experimental): Participants will receive multiple doses of one of different dose levels of VX-708 under fasting condition.
  Interventions: Drug: VX-708
- Part A: Placebo (Placebo Comparator): Participants will receive placebo matched to VX-708.
  Interventions: Drug: Placebo
- Part A: Midazolam With or Without VX-708 (Cohort A4) (Experimental): Participants will receive a single dose of Midazolam with or without VX-708 under fasting condition.
  Interventions: Drug: VX-708; Drug: Midazolam
- Part B: VX-708 With Itraconazole (Experimental): Participants will receive a single dose of VX-708 in treatment period 1, followed by itraconazole, which will be dosed daily with a single dose of VX-708 administered in treatment period 2 under fasting conditions. A washout period of 6 days will be maintained between the 2 treatment periods.
  Interventions: Drug: VX-708; Drug: Itraconazole

INTERVENTIONS:
Drug: VX-708 — Solution for intravenous (IV) administration.
  Arms: Part A: Midazolam With or Without VX-708 (Cohort A4); Part A: VX-708 (Cohort A1-A3); Part B: VX-708 With Itraconazole
Drug: Itraconazole — Solution for oral administration.
  Arms: Part B: VX-708 With Itraconazole
Drug: Midazolam — Solution for oral administration.
  Arms: Part A: Midazolam With or Without VX-708 (Cohort A4)
Drug: Placebo — Placebo matched to VX-708 for IV administration.
  Arms: Part A: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and pharmacodynamics of multiple ascending doses of VX-708 in healthy participants

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female of non-childbearing potential are eligible
* Body mass index (BMI) of 18.0 to 32.0 kilograms per meter square (kg/m^2)
* A total body weight greater than (>) 50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness within 14 days before the first dose of study drug
* History of cardiac dysrhythmias
* Part A Cohorts with Midazolam DDI Evaluation (Cohort A4) Only

  * Hypersensitivity to midazolam or benzodiazepines
* Part A Cohorts with CSF Sampling (Cohorts A2 and A3) Only

  * Hypersensitivity to local anesthetic for lumbar puncture
  * History of conditions leading to increased intracranial pressure (e.g., brain tumor, idiopathic intracranial hypertension, venous sinus thrombosis)
* Part B Only

  * Hypersensitivity to itraconazole

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 30
Part A: Safety and Tolerability as Assessed by Number of Participants With Clinically Meaningful Findings in Columbia Suicide Severity Rating Scale (C-SSRS) Responses | Day 1 up to Day 30
Part A: Continuous Pulse Oximetry Monitoring as assessed by oxygen saturation for Cohort A4 | Pre-dose up to 6 hours Post-dose
Part A: Infusion Nurses Society (INS) Visual Infusion Phlebitis (VIP) Score Monitoring | Day 1 up to Day 30
Part B: Area Under the Plasma Concentration Versus Time Curve from the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-708 in the Absence or Presence of Itraconazole | Day 1 up to Day 16

SECONDARY OUTCOMES:
Part A: Area Under the Plasma Concentration Versus Time Curve from the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-708 | Day 1 up to Day 14
Part A: Area Under the Concentration Versus Time Curve from the Time of Dosing Extrapolated to Infinity (AUC0-inf) of Midazolam and 1-hydroxy-midazolam in the Absence or Presence of VX-708 (Cohort A4) | Day 1 up to Day 14
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 32
Part B: Infusion Nurses Society (INS) Visual Infusion Phlebitis (VIP) Score | Day 1 up to Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion - Tempe, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing